CLINICAL TRIAL: NCT05949476
Title: Influence of Ozone Therapy on Postoperative Pain Relief in the Surgical Treatment of Lower Third Molars: Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera Ordine Mauriziano di Torino (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: OZONOTERAPIA
Record Dates: First submitted 2023-07-10; First posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Extraction of the Lower Third Molars

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): extraction of the lower third molar will be performed according to the standard protocols of the structure
- Trial Group (Experimental): In this group ozone will be used, in two formulations: gaseous, injected into the site of the pre- and post-surgery operation, and topical, in the form of a gel, applied at the end of the operation and for home use according to the therapeutic scheme prescribed at the time of resignation
  Interventions: Other: ozone therapy

INTERVENTIONS:
Other: ozone therapy — Ozone in the gaseous state produced by a machine at concentrations for medical use (sssssssssss9) injected after anesthesia in the surgery site and in the post-extraction alveolus after suture.
  * Topical ozone in the form of a gel (indicate the brand) to be applied to the post-surgical site 2 times a day for 7 days.
  Arms: Trial Group

SUMMARY:
Patients will undergo a split-mouth protocol which includes:

a control group: in which the extraction of the lower third molar will be performed according to the standard protocols of the structure.

A study group: in which ozone will be used in addition, in two formulations: gaseous, injected into the site of the pre- and post-surgery operation, and topical, in the form of a gel, applied at the end of the operation and for home use according to therapeutic scheme prescribed at the time of discharge.

Primary objective: To evaluate whether the use of ozone in patients undergoing extraction of impacted third molars reduces post-operative pain 7 days after surgery.

Secondary objectives:

* Evaluate the functional limitation in opening the mouth (trismus) 7 days after surgery.
* Evaluate if there is a reduced intake of analgesic drugs in the 7 days following the operation.
* Evaluate the perceived quality of life in the 7 days following the intervention.

DETAILED DESCRIPTION:
Patients will undergo a split-mouth protocol which includes:

a control group: in which the extraction of the lower third molar will be performed according to the standard protocols of the structure.

A study group: in which ozone will be used in addition, in two formulations: gaseous, injected into the site of the pre- and post-surgery operation, and topical, in the form of a gel, applied at the end of the operation and for home use according to therapeutic scheme prescribed at the time of discharge.

Primary objective: To evaluate whether the use of ozone in patients undergoing extraction of impacted third molars reduces post-operative pain 7 days after surgery.

Secondary objectives:

* Evaluate the functional limitation in opening the mouth (trismus) 7 days after surgery.
* Evaluate if there is a reduced intake of analgesic drugs in the 7 days following the operation.
* Evaluate the perceived quality of life in the 7 days following the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Lower third molars included
* Pell-Gregory Class II-B
* Absence of systemic diseases

Exclusion Criteria:

* Hyperthyroidism;
* G6PHD (glucose 6 phosphate dehydrogenase) deficiency;
* Anemia
* Myasthenia
* Pregnancy and breastfeeding
* Allergy to ozone
* Local infections

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Estimated)
Dates: Start 2022-07-19 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-19 (Estimated)

PRIMARY OUTCOMES:
Reduction post operative pain | 7 days
  Evaluate whether the use of ozone in patients undergoing extraction of impacted third molars reduces post-operative pain 7 days after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- A.O. Ordine Mauriziano, Torino, Italy

REFERENCES:
- [Derived] Guaschino L, Vanzanelli A, Babando P, Ricotti A, Ramieri GA, Roccuzzo A, Appendino P. Effect of ozone therapy on post-operative pain following mandibular third molar surgical extraction: a split-mouth randomized clinical trial. Clin Oral Investig. 2025 Dec 9;30(1):2. doi: 10.1007/s00784-025-06681-y. PMID 41361069